CLINICAL TRIAL: NCT04887519
Title: Post Authorization Study to Monitor Efficacy, Effectiveness and Safety of Brigatinib (Alunbrig®) in Anaplastic Lymphoma Kinase (ALK) Positive Metastatic Non Small Cell Lung Cancer (NSCLC) in Argentina
Brief Title: A Study of Brigatinib to Treat Adults With Anaplastic Lymphoma Kinase (ALK) Positive Metastatic Non Small Cell Lung Cancer (NSCLC)
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Brigatinib-5008
Record Dates: First submitted 2021-05-13; First posted 2021-05-14 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Anaplastic Lymphoma Kinase
Keywords: Drug Therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Participants: Participants with advanced or metastatic ALK positive NSCLC who have been prescribed with brigatinib in real-world will be observed both prospectively and/or retrospectively at the local clinical practice setting and data will be taken from medical records of the routine visit after every 12 weeks from the start of treatment up to 24 weeks of follow up or death or cancer progression or treatment discontinuation, whichever occurs first.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is a non-interventional study.

SUMMARY:
The aims of the study are to assess the safety profile of brigatinib and the clinical response rates in adults with Anaplastic Lymphoma Kinase (ALK)-Positive Metastatic Non Small Cell Lung Cancer (NSCLC). Treatment with brigatinib and follow-up will be according to routine clinical practice.

Study doctors will review the participants' medical records at the start of the study, then at 12 and 24 weeks after treatment starts.

DETAILED DESCRIPTION:
This is a prospective, observational post-marketing surveillance study of brigatinib in participants with advanced or metastatic NSCLC. This study will assess the safety, efficacy and effectiveness of brigatinib for its approved indications in a routine clinical practice setting under real world use.

The study will enroll approximately 37 participants. The data will be collected both prospectively and/or retrospectively at the specialized centers and outpatient oncology clinics and will be recorded by the investigator in the electronic Case Report Form (eCRF) based on the routine medical care data that is collected in the medical records. All the participants will be assigned to a single observational cohort:

• All Participants

This multi-center study will be conducted in Argentina. The overall duration of the study will be approximately 52 weeks. Data collection will be based on routine visit after every 12 weeks from the start of treatment up to 24 weeks of follow up or death or cancer progression or treatment discontinuation, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. With either a diagnosis of ALK positive metastatic NSCLC previously treated with crizotinib OR a diagnosis of ALK positive metastatic NSCLC previously not treated with an ALK inhibitor. Have received at least one dose of brigatinib according to approved indications.

Exclusion Criteria:

Note: There are no specific exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with a diagnosis of ALK positive metastatic NSCLC that are treated with brigatinib.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2020-12-30 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants Reporting One or More Adverse Events (AEs) of Special Interest | Up to 24 week
  AEs of special interest includes Pneumonitis, interstitial lung disease, including early onset pulmonary events or symptoms; Hypertension; Bradycardia; Drug interactions with strong or moderate CYP3A inhibitors and inducers; hepatic toxicity; Myopathy, including elevation of creatine phosphokinase rhabdomyolysis and cardiomyopathy; Pancreatitis including elevation of lipase and amylase; Macular degeneration, retinopathy and visual disturbances and Embryo-fetal toxicity.
Number of Participants Reporting One or More AEs | Up to 24 week
Number of Participants Reporting One or More Serious Adverse Events (SAEs) | Up to 24 week
Number of Participants Reporting One or More Non-serious Adverse Events (Non-SAEs) | Up to 24 week

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 24 week
  ORR will be evaluated by investigators according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. ORR is defined as the percentage of participants who achieved a best response of a complete response (CR) or partial response (PR). CR: defined as disappearance of all target lesions, non-target lesions, no new lesions, and normalization of tumor marker level. PR: defined as at least a 30 percent (%) decrease in the sum of diameters of target lesions, no progression in non-target lesion, and no new lesions.
Central Nervous System Objective Response Rate (CNS-ORR) | Up to 24 week
  CNS-ORR will be evaluated by the investigator judgement based on usual clinical practice guided by RECIST version1.1 in all participants with evaluable CNS metastases.
Progression-Free Survival (PFS) | From first administration of study drug to the date of disease progression or death due to any cause (up to 24 week)
  PFS will be evaluated by treating physicians according to RECIST version 1.1. PFS is defined as the time from the date of randomization to the date of first documentation of progressive disease or death due to any cause, whichever occurs first.
Overall Survival (OS) | From first administration of study drug to death (up to 24 week)
  OS is defined as the time interval from the date of the first dose of the study treatment until death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- IC Projects, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Martin C, Malcervelli GI, Martinengo GL, Levit P, Servienti P, Malaver E, Brion L, Patronella V, Zumarraga A, Zarba J. Safety and Effectiveness of Brigatinib in Anaplastic Lymphoma Kinase (ALK) Positive Metastatic Non-Small Cell Lung Cancer (NSCLC) in Argentina: A Post-Marketing Surveillance Study. Drugs Real World Outcomes. 2025 Jun;12(2):227-235. doi: 10.1007/s40801-025-00484-z. Epub 2025 Feb 26. PMID 40011377
- See also: Related Info — https://clinicaltrials.takeda.com/study-detail/60a4dea31f1122001e30a7c9